CLINICAL TRIAL: NCT06784674
Title: Diabetes Prediction During Pregnancy Using Pancreas MRI
Brief Title: Maternal Abdominal Morphology Assessment
Acronym: MAMA
Status: Recruiting | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, John Virostko, John Virostko, Associate Professor, Department of Diagnostic Medicine, University of Texas at Austin
Other Study IDs: STUDY00005491
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Infant Development; Pancreas; Diabetes
Keywords: Pregnancy; Pancreas; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood samples will be collected at study visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MAMA Study Participants: Approximately 87 pregnant women, aged 18-54, living in the Greater Austin area, will participate in the MAMA study. The MAMA study is an observational study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
Previous studies have shown that pancreas size tends to be smaller in individuals with diabetes compared to those without diabetes. The investigators have recently found that pancreas size increases during pregnancy. The MAMA study aims to examine changes in the pancreas that occur during pregnancy, in both pregnant mothers and their babies, and find out how they are affected by maternal diabetes.

The MAMA study is a prospective cohort study that will follow women and their babies through pregnancy and one year postpartum. Women aged 18-54, who are under 14 weeks pregnant are being recruited to participate in the MAMA study.

DETAILED DESCRIPTION:
As pancreas size is thought to reflect pancreatic insulin production and/or islet mass, monitoring pancreas size during and after pregnancy may advance the investigators' understanding of gestational diabetes mellitus (GDM) incidence and progression. Information on pancreas size changes during pregnancy, typical fetal pancreatic development, the relationship between pancreas size and GDM risk, and the relationship between pancreas size and neonatal hypoglycemia are largely unknown. Through this project, magnetic resonance imaging (MRI) will be used to measure changes in pancreas size during pregnancy and the effect of maternal diabetes on these measures.

This prospective cohort study is observational and will include up to 87 pregnant women who are between 18-54 years old. Study visits will take place at approximately 15-18 weeks gestation, 24-28 weeks gestation, 34-38 weeks gestation, and 1 year-1 year and 2 months postpartum. At each study visit, participants will self-report their height and weight, have their blood pressure measured, have their blood drawn, have an HbA1c finger stick test, participate in oral glucose tolerance testing (OGTT), complete an MRI scan, and undergo continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, with a singleton gestation
* Age 18 - 54 years at screening
* Gestational age < 14 weeks
* Willing to commit to 1 year postpartum follow up
* Planning to remain in geographical vicinity of Austin for 1 year after delivery

Exclusion Criteria:

* Presence of any mechanically or magnetically activated implants
* Claustrophobia
* Other contraindication for MRI
* BMI ≥ 38.0 or maximum width less than 48 cm (necessary to fit within the MRI field of view)

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators intend to enroll 87 total participants. The study population will consist of women who are under 14 weeks pregnant with a singleton gestation, aged 18-54, living in the Greater Austin Area.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Maternal Pancreatic Volume | 15-18 weeks gestation, 24-28 weeks gestation, and 34-38 weeks gestation as well as 1 year-1 year and 2 months postpartum.
  Maternal pancreatic volume will be measured at each study visit. MRI will be utilized to determine maternal pancreatic volume in cm^3.
Fetal Pancreatic Volume | 15-18 weeks gestation, 24-28 weeks gestation, and 34-38 weeks gestation.
  Fetal pancreatic volume will be measured at each study visit. MRI will be utilized to determine fetal pancreatic volume in utero in cm^3. Fetal pancreatic volume will not be ascertained at the final study visit.

SECONDARY OUTCOMES:
Plasma Insulin | 15-18 weeks gestation, 24-28 weeks gestation, and 34-38 weeks gestation as well as 1 year-1 year and 2 months postpartum.
  Plasma Insulin values (µU/mL or pmol/L) measured via blood draw will be utilized to calculate Glycemic Control and Insulin Sensitivity.
Plasma Glucose | 15-18 weeks gestation, 24-28 weeks gestation, and 34-38 weeks gestation as well as 1 year-1 year and 2 months postpartum.
  Plasma Insulin values (mg/dL or mmol/L) measured via blood draw will be utilized to calculate Glycemic Control and Insulin Sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Virostko, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Dell Medical School Health Discovery Building, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No